CLINICAL TRIAL: NCT03370887
Title: A Randomized, Double-blind, Placebo-controlled, Multi-centre, Sequential Design, Phase IIa Study to Evaluate Safety and Tolerability of Epicardial Injections of AZD8601 During Coronary Artery Bypass Grafting Surgery
Brief Title: AZD8601 Study in CABG Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: D9150C00003
Record Dates: First submitted 2017-11-16; First posted 2017-12-13 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose AZD8601 (3 mg) (Experimental): 8 patients will be randomised to receive 3 mg AZD8601
  Interventions: Drug: AZD8601
- High dose AZD8601 (30 mg) (Experimental): 8 patients will be randomised to receive 30 mg AZD8601
  Interventions: Drug: AZD8601
- Placebo (Placebo Comparator): 8 patients will be randomised to receive placebo injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8601 — AZD8601 solution for injection, 0,5 mg/mL and 5 mg/mL will be given as 30 injections of 0.1 mg (3 mg per patient), or 1 mg (30 mg per patient) respectively on a single occasion
  Arms: High dose AZD8601 (30 mg); Low dose AZD8601 (3 mg)
Drug: Placebo — Placebo for AZ8601 injection for solution will be given as 30 injections per patient on a single occasion
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, sequential design, multicentre study in patients with moderately impaired systolic function undergoing CABG surgery. Twenty four (24) patients scheduled for elective bypass surgery will be randomized (up to approximately 33 patients if replacements are needed). The objective is to investigate safety and tolerability of AZD8601 following epicardial injection in patients undergoing Coronary Artery Bypass Grafting (CABG) surgery with moderately impaired systolic function. At Visit 3 patients will receive either AZD8601 or placebo as epicardial injections and will then be followed up at 14 days (telephone visit) and 1, 3 and 6 months (on-site) post-surgery.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study patients should fulfil the following criteria at Visit 1 and/or 2:

1. Provision of signed and dated informed consent prior to any study specific procedures

Males and females:

1. Males must be surgically sterile or using an acceptable method of contraception
2. Females must be of non-childbearing potential confirmed at screening by fulfilling one of the following criteria a) postmenopausal defined as amenorrhoea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the postmenopausal range, b) documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation 3. Age >18 years 4. Indication for elective CABG surgery enrolled at least 15 days before the planned surgery 5. Moderately reduced global LVEF at rest (30% ≤ LVEF ≤ 50%) from medical records 6. If patient is on statin, ACE inhibitor/ARB, and/or beta-blocker, the dose should be stable at least 2 weeks prior to Visit 1 7. Patients who are blood donors should not donate blood during the study and for 3 months following their last dose of AZD8601.

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site) 2. Previous randomisation in the present study 3. Participation in another clinical study with an investigational product during the last 3 months 4. BMI > 35 kg/m2 OR poor image window for echocardiography 5. Need for CABG emergency operation. (Emergency operation is defined as significant symptom status worsening in CAD, such as crescendo angina, unstable angina or ACS requiring rescheduling the revascularization. CAD should be stable at least 3 months prior to Visit 3.) 6. History of ventricular arrhythmia (≥ Lown III) without Implantable Cardiac Defibrillator (ICD) History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study 8. Severe co-morbidities that can interfere with the execution of the study, interpretation of study results or affect the safety of the patient, in judgement of the investigator 9. eGFR ≤ 30 mL/min (derived from creatinine clearance, calculated by local lab) 10. For CFVR (Visit 1) and sMBF (Visit 2) measurement:

* Known severe adverse reactions to adenosine
* Known elevated intracranial pressure
* AV block ≥ second degree and/or sick sinus syndrome in patient without pacemaker
* Heart rate < 40 bpm (ECG verified)
* Systolic blood pressure < 90 mmHg
* Asthma or COPD with strong reactive component in judgement of investigator
* Treatment with dipyridamole (e.g. Persantin or Asasantin), theophyllamine or fluvoxamine that cannot be paused 11. Inability to comply with the protocol 12. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity to drugs with a similar chemical structure or class as study drugs 13. Patients unable to give their consent or communicate reliably with the investigator or vulnerable patients e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order 14. Positive hepatitis C antibody hepatitis B virus surface antigen or hepatitis B virus core antibody or human immunodeficiency virus, at Visit 1 15. Known history of drug or alcohol abuse 16. Any concomitant medications that are known to be associated with Torsades de Pointes 17. History of QT prolongation associated with other medications that required discontinuation of that medication 18. Congenital long QT syndrome 19. History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTCAE Grade 3).

  20. Current atrial fibrillation as well as paroxysmal atrial fibrillation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vesa Anttila, MD, PhD, Principal Investigator — Heart Center, Turku University, Finland
Locations (9):
- Research Site, New Haven, Connecticut, United States
- Finland (3):
  - Research Site, Kuopio
  - Research Site, Tampere
  - Research Site, Turku
- Research Site, München, Germany
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Groningen
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Anttila V, Saraste A, Knuuti J, Hedman M, Jaakkola P, Laugwitz KL, Krane M, Jeppsson A, Sillanmaki S, Rosenmeier J, Zingmark P, Rudvik A, Garkaviy P, Watson C, Pangalos MN, Chien KR, Fritsche-Danielson R, Collen A, Gan LM. Direct intramyocardial injection of VEGF mRNA in patients undergoing coronary artery bypass grafting. Mol Ther. 2023 Mar 1;31(3):866-874. doi: 10.1016/j.ymthe.2022.11.017. Epub 2022 Dec 17. PMID 36528793
- [Derived] Anttila V, Saraste A, Knuuti J, Jaakkola P, Hedman M, Svedlund S, Lagerstrom-Fermer M, Kjaer M, Jeppsson A, Gan LM. Synthetic mRNA Encoding VEGF-A in Patients Undergoing Coronary Artery Bypass Grafting: Design of a Phase 2a Clinical Trial. Mol Ther Methods Clin Dev. 2020 Jun 1;18:464-472. doi: 10.1016/j.omtm.2020.05.030. eCollection 2020 Sep 11. PMID 32728595
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9150C00003&attachmentIdentifier=5b906a96-c6ba-4875-a07c-483c962a67f7&fileName=CSP_redacted.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9150C00003&attachmentIdentifier=973817b6-2b81-463b-911d-85e1e0dc6df6&fileName=SAP_redacted.pdf&versionIdentifier=
- See also: CSR synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9150C00003&attachmentIdentifier=00b9c773-8ec2-4f49-a95b-0dd4b2be164c&fileName=CSR_synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 4 clinical research centers in Finland and Germany First subject enrolled (First subject first visit/first consent signed date): 2018. Last subject last visit: 2021.
Pre-assignment Details: The study was to include two dose cohorts, which were to receive a total dose of 3 or 30 mg ofAZD8601. However, due to low recruitment levels, only 7 participants receiving a total dose of 3 mg AZD8601 and 4 participants receiving placebo completed dosing, according to the randomisation scheme
Groups:
- AZD8601 3mg: AZD8601 3mg
- Placebo: Placebo
Period: Overall Study
Arm/Group | AZD8601 3mg | Placebo
Started | 7 | 4
Completed | 7 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD8601 3mg | Placebo | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.3 (5.8) | 67.8 (10.8) | 68.1 (7.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 7 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Time Frame: From baseline to end of follow up at 6 months
Measure: Count of Participants; unit: Participants
Groups:
- AZD8601 3 mg: AZD8601 3 mg
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 7 | 4
Participants | 7 | 4

2. Primary Outcome: Pulse Rate (Vital Sign)
Time Frame: From baseline to end of follow up at 6 months
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 7 | 4
beats/min
  Baseline | 63.1 (10.42) | 62.6 (6.04)
  Day 1 | 81.3 (7.38) | 75.2 (4.20)
  Day 2 | 85.2 (5.54) | 81.1 (7.01)
  Day 3 | 83.6 (8.38) | 82.4 (6.80)
  Day 4 | 81.9 (14.54) | 75.3 (7.63)
  Visit 5 (Day 30) | 74.3 (13.33) | 65.5 (6.81)
  Visit 6 (Day 91) | 66.9 (15.05) | 70.8 (7.18)
  Visit 7 (Day 182) | 63.6 (15.62) | 61.0 (2.16)

3. Primary Outcome: Number of Subjects With an ECG Determined to be Abnormal and Clinically Significant
Time Frame: From baseline to end of follow up at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 7 | 4
Participants
  Baseline | 0 | 0
  End of treatment | 1 | 0

4. Primary Outcome: Number of Subjects With High Values of Leukocytes, Particle Concentration
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 6 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 3 | 1

5. Primary Outcome: Oxygen Saturation (Vital Sign)
Time Frame: From baseline to end of follow up at 6 months
Population: No SD calculated when only one subject in group
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 7 | 4
Percent
  Baseline: number analyzed (Participants) | 1 | 1
  Baseline | 96.0 | 100.0
  Day 1 | 97.6 (4.46) | 99.3 (0.80)
  Day 2: number analyzed (Participants) | 6 | 4
  Day 2 | 97.7 (1.68) | 97.4 (2.42)
  Day 3: number analyzed (Participants) | 6 | 4
  Day 3 | 95.6 (2.14) | 96.6 (3.60)
  Day 4: number analyzed (Participants) | 6 | 4
  Day 4 | 95.7 (1.85) | 95.8 (3.74)

6. Primary Outcome: Systolic Blood Pressure (Vital Sign)
Time Frame: From baseline to end of follow up at 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 7 | 4
mmHg
  Baseline | 141.1 (24.42) | 141.7 (23.32)
  Day 1 | 113.5 (5.67) | 116.8 (12.53)
  Day 2 | 118.1 (11.98) | 104.8 (4.39)
  Day 3 | 118.5 (8.04) | 100.8 (10.82)
  Day 4 | 129.1 (16.63) | 109.0 (6.48)
  Visit 5 (Day 30) | 135.9 (17.56) | 134.5 (29.49)
  Visit 6 (Day 91) | 146.3 (11.76) | 163.0 (35.39)
  Visit 7 (Day 182) | 142.3 (13.00) | 147.3 (34.07)

7. Primary Outcome: Number of Subjects With High Values of Erythrocytes, Particle Concentration
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 5 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 0

8. Primary Outcome: Diastolic Blood Pressure (Vital Sign)
Time Frame: From baseline to end of follow up at 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 7 | 4
mmHg
  Baseline | 82.1 (17.95) | 74.5 (23.57)
  Day 1 | 59.2 (6.52) | 62.0 (7.63)
  Day 2 | 59.2 (10.62) | 58.0 (5.12)
  Day 3 | 63.7 (8.64) | 56.9 (2.83)
  Day 4 | 73.7 (11.07) | 66.8 (5.91)
  Visit 5 (Day 30) | 78.1 (10.16) | 83.5 (14.55)
  Visit 6 (Day 91) | 80.0 (7.09) | 93.8 (16.62)
  Visit 7 (Day 182) | 79.4 (8.06) | 83.5 (19.60)

9. Primary Outcome: Number of Subjects With High Values of Erythrocyte, Volume Fraction
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 6 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 0

10. Primary Outcome: Number of Subjects With High Values of Erythrocytes, Mean Cell Volume
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 6 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 1 | 0

11. Primary Outcome: Number of Subjects With High Values of Hemoglobin
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 6 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 0

12. Primary Outcome: Number of Subjects With High Values of Neutrophils
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 5 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 2 | 0

13. Primary Outcome: Number of Subjects With High Values of Lymphocytes
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 5 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 0

14. Primary Outcome: Number of Subjects With High Values of Monocytes
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 5 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 1

15. Primary Outcome: Number of Subjects With High Values of Eosinophils
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 5 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 0

16. Primary Outcome: Number of Subjects With High Values of Basophils
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 5 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 0

17. Primary Outcome: Number of Subjects With High Values of Platelets
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 6 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 0

18. Primary Outcome: Number of Subjects With High Values of Reticulocytes
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 5 | 2
Number of subjects
  Baseline | 1 | 1
  Maximum value during treatment | 1 | 0

19. Primary Outcome: Number of Subjects With High Values of Prothrombin Complex INR
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 4 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 0

20. Primary Outcome: Number of Subjects With High Values of Activated Partial Thromboplastin Time
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 4 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 0

21. Primary Outcome: Number of Subjects With High Values of Fibrinogen
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 3 | 3
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 3 | 2

22. Primary Outcome: Number of Subjects With High Values of Sodium
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 6 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 0

23. Primary Outcome: Number of Subjects With High Values of Potassium
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 6 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 0

24. Primary Outcome: Number of Subjects With High Values of Urea
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 4 | 4
Number of subjects
  Baseline | 0 | 1
  Maximum value during treatment | 0 | 0

25. Primary Outcome: Number of Subjects With High Values of Creatinine
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 5 | 4
Number of subjects
  Baseline | 1 | 1
  Maximum value during treatment | 1 | 1

26. Primary Outcome: Number of Subjects With High Values of Albumin
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 5 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 0

27. Primary Outcome: Number of Subjects With High Values of Calcium
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 5 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 0

28. Primary Outcome: Number of Subjects With High Values of Phosphate
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 4 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 0 | 0

29. Primary Outcome: Number of Subjects With High Values of Alkaline Phosphatase
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 5 | 4
Number of subjects
  Baseline | 0 | 1
  Maximum value during treatment | 0 | 1

30. Primary Outcome: Number of Subjects With High Values of Alanine Aminotransferase
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 5 | 4
Number of subjects
  Baseline | 0 | 1
  Maximum value during treatment | 0 | 0

31. Primary Outcome: Number of Subjects With High Values of Aspartate Aminotransferase
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 5 | 4
Number of subjects
  Baseline | 1 | 1
  Maximum value during treatment | 0 | 1

32. Primary Outcome: Number of Subjects With High Values of Bilirubin, Total
Description: Values are classified as high if they are above the normal reference range, based on local lab reference ranges.
Time Frame: From baseline to end of follow up at 6 months
Population: For some participants laboratory analysis have not been made
Measure: Number; unit: Number of subjects
Arm/Group | AZD8601 3 mg | Placebo
Number analyzed (Participants) | 5 | 4
Number of subjects
  Baseline | 0 | 0
  Maximum value during treatment | 1 | 0

ADVERSE EVENTS:
Time Frame: All adverse events are summarized from the dose of IP to the end the follow-up period at 6 months.
Arm/Group | AZD8601 3mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/7 | 1/4
Other Adverse Events (participants affected / at risk) | 7/7 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8601 3mg (N=7) | Placebo (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Incision site impaired healing (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8601 3mg (N=7) | Placebo (N=4)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Embolic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT03370887/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT03370887/SAP_001.pdf